CLINICAL TRIAL: NCT02486575
Title: Comparison of Laparoscopic Simulation Training Between Mentoring and Self-learning Technique
Brief Title: Trial on Laparoscopic Simulation Based on Mentoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Federico Gheza, Research specialist, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TUTOR LAP SYM
Record Dates: First submitted 2014-01-24; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Performance of Wrong Procedure (Operation)
Keywords: Residents; Training; simulation; mentoring; proctor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-learning (Other): Residents training alone with pre-recorded instructions. No tutor intervention, only self-learning training Intervention Type: Behavioral (video-based and instruction based learning)
  Interventions: Other: Self-learning
- Mentoring (Other): Residents training with a mentor, giving tailored instruction to each of them and correction to wrong behaviours.
  Intervention Type: Behavioral (tutored learning)
  Interventions: Other: Mentoring

INTERVENTIONS:
Other: Self-learning — Every resident will train following the video instruction included in the FLS course material and related written instruction only
  Arms: self-learning
Other: Mentoring — A tutor will follow each resident during learning, giving instruction, examples and any kind of suggestions.
  Arms: Mentoring

SUMMARY:
More than 50 residents in surgical specialities (OB&G, General surgery and Urology) from a single university in Italy will be randomized into two groups, after a stratification based on residency year and laparoscopic/simulator experience. The first one will train to FLS (fundamentals of laparoscopic surgery) following pre-recorded instruction from course materials; the second one will be mentored by a proctor in single training section. The aim is to evaluate the best way to train residents applying for the very first time in an extensive way the "fundamentals of laparoscopic surgery" program in an Italian Institution.

DETAILED DESCRIPTION:
A complete 5-skills based FLS (fundamentals of laparoscopic surgery) curriculum is proposed to each resident enrolled in the trial. The first group trains with videos and written instructions, without any kind of support from a tutor. The second group is aided by a tutor, receiving tailored teaching and mentoring.

The primary goal was to asses the impact of tutoring in Passing the FLS examination at the end of a 3-months training: the outcome is the dichotomous PASS/DON'T PASS THE EXAM. At the same time the investigators assess the performance to record and evaluate any differences in groups and subgroups (year of residency, gender, specialty, etc.).

The evaluation was based on FLS program standards, recording time and penalties.

The training and evaluation setting was created to exactly reproduce the FLS one, mostly using the FLS material itself, or using FLS admitted/compatible instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Residents in surgical specialities at University of Brescia

Exclusion Criteria:

* Residents not available for the training (outside the Country, not interested, etc.)

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Performance at FLS (fundamentals of laparoscopic surgery) test at the end of training as defined from SAGES | 2 months to compleete the training
  2 months for the training and final evaluation in 2 weeks. Parameters evaluated during the final test are as defined by SAGES at "http://www.flsprogram.org" in the "manual skills" module.

CONTACTS AND LOCATIONS:
Overall Officials: Nazario Portolani, MD, Study Director — Università degli Studi di Brescia

REFERENCES:
- [Derived] Gheza F, Raimondi P, Solaini L, Coccolini F, Baiocchi GL, Portolani N, Tiberio GAM. Impact of one-to-one tutoring on fundamentals of laparoscopic surgery (FLS) passing rate in a single center experience outside the United States: a randomized controlled trial. Surg Endosc. 2018 Nov;32(11):4428-4435. doi: 10.1007/s00464-018-6185-1. Epub 2018 Apr 11. PMID 29644465